CLINICAL TRIAL: NCT04366375
Title: Comparison of the Tissue Trauma Markers Following Total Laparoscopic Hysterectomy vs Total Abdominal Hysterectomy
Brief Title: Pentraxin-3 in Hysterectomy Patients
Status: Completed | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Burak Sezgin, Principal Investigator, Muğla Sıtkı Koçman University
Other Study IDs: 19.03.15-58-56
Record Dates: First submitted 2020-04-25; First posted 2020-04-28 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Laparoscopic Hysterectomy; Abdominal Hysterectomy
Keywords: Pentraxin-3; tissue trauma; hysterectomy; neutrophil to lymphocyte ratio

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum blood samples for each participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TLH+BSO: Total Laparoscopic Hysterectomy + Bilateral Salpingo-Oophorectomy N=20
  Interventions: Diagnostic Test: PTX-3
- TAH + BSO: Total Abdominal Hysterectomy + BSO N=20
  Interventions: Diagnostic Test: PTX-3

INTERVENTIONS:
Diagnostic Test: PTX-3 — Pentraxin-3 ng/mL PTX-3 levels were measured using human PTX3 ELISA Kit 96 Tests/Box (Cat. No: CK-E90303) (Hangzhou Eastbiopharm Co.,Ltd., PRC) read by a ELISA device matching with the kit. For the purpose of measurement, microplate washer RT 2600 device and Rayto microplate reader RT 2100C device were used.

SUMMARY:
Comparison of the Tissue Trauma Markers Following Total Laparoscopic Hysterectomy vs Total Abdominal Hysterectomy

DETAILED DESCRIPTION:
Acute trauma and major surgeries activate a series of cascades to evoke systemic inflammatory response. The magnitude of the resulting inflammatory response is proportional to the severity of the tissue trauma. Abdominal or laparoscopic technique is widely used for the purpose of hysterectomy surgery. It is crucial for many aspects to compare these two techniques of hysterectomy in terms of the surgery-induced trauma.

In this study, the severity of the inflammatory response resulting from the tissue trauma due to the techniques of TLH+BSO and TAH+BSO applied in our department were compared based on the PTX-3 molecule.

ELIGIBILITY:
Inclusion Criteria:

·TLH+BSO patients and TAH+BSO patients

Exclusion Criteria:

* History of a chronic disease (coronary artery disease, diabetes mellitus, hypertension, coronary liver failures, chronic kidney disease, chronic respiratory diseases, connective tissue disorders) which may affect levels of PTX-3 and other inflammatory markers.
* Prior surgery due to malignancy.
* History of an intra-abdominal surgery, except for cesarean section.
* History of any disease which may lead to intra-abdominal adhesions (endometriosis, past pelvic infection).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — TLH+BSO and TAH+BSO applied patients
Study Population: A total of 40 patients, composed of 20 TLH+BSO patients and 20 TAH+BSO patients were included into the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-01-13 (Actual); Primary Completion 2015-12-07 (Actual); Study Completion 2015-12-07 (Actual)

PRIMARY OUTCOMES:
Pentraxin-3 level | Before 24 hours preoperatively and upto 24 hours postoperatively
  Pentraxin-3 ng/mL

SECONDARY OUTCOMES:
(NLR) | Up to 24 hours postoperative
  neutrophile/lymphocyte ratio

CONTACTS AND LOCATIONS:
Overall Officials: Burak SEZGİN, Dr, Principal Investigator — Mugla Sıtkı Kocman University Faculty of Medicine

IPD SHARING:
Plan to Share IPD: Undecided
undecided